CLINICAL TRIAL: NCT05472493
Title: Nuclear Imaging for Subtype Diagnosis of Primary Aldosteronism
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REB22-0772
Record Dates: First submitted 2022-07-18; First posted 2022-07-25 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CETO (Experimental): The consented participants will receive the [18-F] CETO through the IV and a PET/CT scan afterwards.
  Interventions: Biological: [18-F]CETO

INTERVENTIONS:
Biological: [18-F]CETO — PET/CT will be performed; Non-contrast CT images will be acquired over the adrenals (slice width, ~3 mm). CETO (~2.5 MBq/kg; up to 365 MBq +/- 20%) will be administered as a single dose intravenously and dynamic PET images will be acquired from ~0-90 minutes.

SUMMARY:
This study is to evaluate the accuracy of a novel radiopharmaceutical tracer, para-chloro-2-[18F]fluoroethyl etomidate (CETO), used with positron emission tomography (PET) and computed tomography (CT), as a way to subtype unilateral vs. bilateral forms of Primary Aldosteronism, compared to AVS as a reference gold standard.

DETAILED DESCRIPTION:
This is a phase II study (with targeted recruitment of 30 participants) designed to evaluate the accuracy of a novel radiopharmaceutical tracer, para-chloro-2-[18F]fluoroethyl etomidate (CETO), used with positron emission tomography (PET) and computed tomography (CT), as a way to subtype unilateral vs. bilateral forms of Primary Aldosteronism, compared to AVS as a reference gold standard. Subjects consenting to study participation will receive the [18-F] CETO followed by the PET/CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with hypertension
* Individuals with an elevated screening adrenal renin ratio (ARR)
* Individuals with or without spontaneous or diuretic-induced hypokalemia, and/ or plus a discrete adrenal nodule or nodules (1 cm or greater) with concordant lateralization on AVS.

Exclusion Criteria:

* Individuals with chronic kidney disease (estimated glomerular filtration rate <40 mL/min/1.73m2),
* Individuals with a history of uncontrolled severe hypertension (>180/110 mmHg), severe uncontrolled diabetes, suspected or proven hypercortisolism (e.g., cortisol-secreting adrenal adenoma), or individuals with an anatomical disease of the liver (e.g., hepatic adenoma or focal nodular hyperplasia)
* Allergy to intravenous contrast, coagulopathy, use of chronic corticosteroids.
* Pregnancy, lactation, and pheochromocytoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is diagnostic test accuracy (expressed as sensitivity, specificity, positive predictive value, and negative predictive value) for CETO PET/CT using adrenal vein sampling as a reference standard. | It will be measured using adrenal vein sampling approximately the same time as the CETO PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Leung, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No